CLINICAL TRIAL: NCT07065994
Title: The Effect of Virtual Reality Glasses Application on Pain and Anxiety Levels in Colorectal Surgery Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Tuba Yılmazer, Principal investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: colorectalsurgery
Record Dates: First submitted 2025-06-26; First posted 2025-07-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Surgery; Virtual Reality; Nursing Care; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): All patients in the experimental group will be asked to fill out the "Informed Consent Form" the day before the surgery, and the patients who agree to participate in the study will be asked to fill out the "Patient Introduction Form" and the "State Anxiety Scale" by the researchers.
  The "Simulator Illness Questionnaire" used in the Virtual Reality disease field will be applied to the experimental group to determine their physiological status before the application. Then, a relaxing music-backgrounded video containing nature images will be watched with virtual reality glasses for 10-15 minutes the day before the surgery. Then, the "Simulator Illness Questionnaire" and the "State Anxiety Scale" will be filled out again.
  The "Simulator Illness Questionnaire" will be applied to the patients at the most appropriate time after the surgery, when their vital signs have stabilized and clinical compliance has been achieved, and 2 hours after their transfer from the postoperative care unit to th
  Interventions: Device: Virtual Reality Glasses Application
- Control (No Intervention): All patients in the control group will be given permission with the "Informed Consent Form" the day before the surgery, and the patients who agree to participate in the study will be asked to fill out the "Patient Introduction Form" and the "State Anxiety Scale" by the researchers.
  No intervention will be applied to the control group patients, and the routine practices of the clinic will continue.
  All patients in the experimental and control groups will be assessed for pain with the Visual Analog Scale (VAS) at the 2nd and 4th hours, and the "State Anxiety Scale" will be applied.

INTERVENTIONS:
Device: Virtual Reality Glasses Application — The day before the surgery, you will be shown a video of nature images with relaxing music for 10-15 minutes using virtual reality glasses.
  Arms: Experimental

SUMMARY:
This study aims to determine the effect of virtual reality glasses on pain and anxiety levels in colorectal surgery patients. This study is a single-center, parallel-group, open-label, randomized controlled clinical trial. This study will be conducted with 60 patients who underwent colorectal surgery between August 2025 and December 2025. Participants will be randomized into two groups as the intervention group (n=30) and the control group (n=30).

All patients in the experimental and control groups will be asked to fill out the "Informed Consent Form" the day before the surgery, and the patients who agree to participate in the study will be asked to fill out the "Patient Introduction Form" and the "State Anxiety Scale" by the researchers.

The "Simulator Illness Questionnaire" used in the Virtual Reality disease field will be applied to the experimental group to determine their physiological conditions before the application. Then, a relaxing music-backgrounded video containing images of nature will be watched with virtual reality glasses for 10-15 minutes the day before the surgery. Then, the "Simulator Illness Questionnaire" and the "State Anxiety Scale" will be filled out again.

The "Simulator Illness Questionnaire" will be applied to the patients 2 hours after their transfer from the postoperative care unit to the clinic, which is the most appropriate time after the surgery, when their vital signs have stabilized and clinical compliance has been achieved, and their physiological conditions before the application will be determined. Then, the patients in the experimental group will be asked to watch a relaxing music-backgrounded video containing images of nature for 10-15 minutes with virtual reality glasses. The researcher will perform the video with virtual reality glasses in the patient rooms and beds. Afterwards, the "Simulator Disease Survey" will be repeated. There will be no compelling effect that will negatively affect the health of the patients during the application, and the application will be terminated when the patients feel uncomfortable. A safe environment will be created so that there are no objects around the patients that they can bump into or trip over. A 5-10 minute trial period will be performed at the beginning with the observer and the virtual reality glasses will be applied. The patient will be able to end the study at any time. If the patients use glasses/lenses, compliance will be checked.

No intervention will be applied to the control group patients and the routine practices of the clinic will continue.

All patients in the experimental and control groups will be assessed for pain with the Visual Analog Scale (VAS) at the 2nd and 4th hours and the "State Anxiety Scale" will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older, 65 years of age or younger,
* Who will undergo laparoscopic colorectal surgery,
* Who do not develop any complications during or after the surgical procedure,
* Who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Patients who have not undergone laparoscopic surgery,
* Those who are hemodynamically unstable,
* Those with neurological or psychological problems,
* Those who are transferred to the intensive care unit after surgery,
* Emergency and unplanned cases,
* Those with visual, auditory or systemic disorders,
* Those who have balance problems,
* Those diagnosed with hypertension or hypotension,
* Patients diagnosed with anxiety disorder or epilepsy will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | preoperative, postoperative 2 hours, postoperative 4 hours
  VAS is a scale consisting of 10 cm lines (0-10 cm) used to assess pain. 0 means "no pain" and 10 means "unbearable pain". In this method, the patient is asked to mark the number between these two extreme points and the degree of pain (F. E. Aslan, 2002).
Spielberger State and Trait Anxiety Inventory (STAI) | preoperative, postoperative 2 hours, postoperative 4 hours
  STAI, which is widely used and still valid, was developed by Spielberger, Gorsuch and Lushene in 1970, and its Turkish language and content validity was made by Öner and Le Compte in 1983. It consists of 2 subscales covering 20 statements measuring state and trait anxiety. The State Anxiety Subscale (STAI-S) expresses how an individual feels at a certain moment and under certain conditions; and the Trait Anxiety Subscale (STAI-T) expresses how they generally feel. The inventory is answered through 4-dimensional definitions. The feelings and behaviors expressed in the State Anxiety Subscale items are specified by selecting one of the options "(1) None, (2) Some, (3) A lot and (4) Completely" according to the severity of such experiences. The feelings and behaviors expressed in the Trait Anxiety Subscale items are specified according to their frequency levels; It is expressed as "(1) Almost Never, (2) Sometimes, (3) A Lot of the Time, and (4) Almost Always". High scores from each subsca
Simulator Sickness Questionnaire (SSQ) | preoperative, postoperative 2 hours
  Simulation Sickness Questionnaire (SSQ) is widely used to measure Virtual Reality sickness (Sevinc and Berkman, 2020, Igoshina et al. 2022). Simulator sickness questionnaire consists of 16 questions. These questions are located under 4 components: nausea (N), oculomotor (O), disorientation (D) and weighted total (T). The majority of studies conducted using SSQ reported only the Total Score score (Sevinc, and Berkman, 2020).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)